CLINICAL TRIAL: NCT00953914
Title: Pyridostigmine and Its Effects on Autonomic Modulation in Diabetic Patients With Autonomic Neuropathy
Brief Title: Pyridostigmine and Its Effects on Autonomic Modulation in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Ruy Silveira Moraes Filho, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04471
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Diabetes Complications
Keywords: pyridostigmine; autonomic modulation; diabetes mellitus; heart rate variability
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus | interventions — Pyridostigmine Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pyridostigmine (Experimental)
  Interventions: Drug: Pyridostigmine
- Placebo (Placebo Comparator): If a subject is randomized to placebo, he will receive placebo pills 3 times daily for 1 day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyridostigmine — Pills containing 30 mg of Pyridostigmine will be orally administered 3 times daily for 1 day.
  Arms: Pyridostigmine
Drug: Placebo — If subject is randomized to placebo, placebo pills will give 30 mg orally 3 times daily for 2 days
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine if pyridostigmine bromide improves heart rate variability of type 2 diabetes mellitus subjects with cardiovascular autonomic neuropathy.

DETAILED DESCRIPTION:
The reduced heart rate variability is associated with increased risk of death in patients with diabetes mellitus. Cholinesterase inhibition with pyridostigmine bromide increases heart rate variability in normal individuals and congestive heart failure subjects but its effects on patients with diabetes mellitus is unknown. Based on those evidences, we will test if the short-term administration of pyridostigmine bromide increases heart rate variability in patients with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus

Exclusion Criteria:

* myocardial infarction
* acute ischemic syndromes
* second or third degree atrioventricular block
* active alcoholism
* thyroid dysfunction
* chronic obstructive pulmonary disease
* history of intolerance to pyridostigmine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-03; Primary Completion 2009-07 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
autonomic modulation assessed by heart rate variability | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Ruy S. Moraes, MD, Phd, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Behling A, Moraes RS, Rohde LE, Ferlin EL, Nobrega AC, Ribeiro JP. Cholinergic stimulation with pyridostigmine reduces ventricular arrhythmia and enhances heart rate variability in heart failure. Am Heart J. 2003 Sep;146(3):494-500. doi: 10.1016/S0002-8703(03)00319-3. PMID 12947369